CLINICAL TRIAL: NCT02995057
Title: Safety Demonstration of Microneedle Insertion
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: H14-02324
Record Dates: First submitted 2015-08-26; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Allergic Reaction to Nickel
Keywords: Microneedles; Biocompatibility; Allergy; Metal; Nickel; Contact dermatitis
MeSH Terms: conditions — Hypersensitivity; Dermatitis, Contact

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nickel allergic: Participants have proven nickel allergy
  Interventions: Device: Gold- or silver-coated, or uncoated nickel microneedles

INTERVENTIONS:
Device: Gold- or silver-coated, or uncoated nickel microneedles — The stratum corneum of the participants will be breached with the gold- and silver-coated, or uncoated nickel microneedles.

SUMMARY:
Hypodermic needles are conventionally used to deliver drugs and vaccines into the muscle of humans and animals. Side effects of these needle injections are pain, bleeding, and anxiety in patients. An alternative drug and vaccine delivery method is the use of hollow microneedles, which are sub-millimeter needle-like structures. Microneedles are pain- and bleeding-free, as they do not reach the nerve-endings and blood capillaries in the skin. As a result, they are better received by patients and do not induce needle anxiety. As the investigators' microneedles are made of gold- or silver-coated, as well as uncoated nickel, the purpose of this study is to observe their biocompatibility and inertness.

ELIGIBILITY:
Inclusion Criteria:

* Proven nickel allergy

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 15 subjects will be enrolled in the trial. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be eligible to enroll in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Skin reaction as measured by a contact dermatitis classification system | 7 days
  Allergic patch-test based grading will be done according to the Wilkinson DS et al 1970 reference.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Hafeli, Ph.D., Principal Investigator — Professor
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No